CLINICAL TRIAL: NCT01604525
Title: RealU: Tailored Web and Peer Email Cessation Counseling for College Smokers
Brief Title: Tailored Web and Peer Email Cessation Counseling for College Smokers
Acronym: RealU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Lawrence C. An, Associate Professor of Internal Medicine, Medical School, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01HL089491 (NIH)
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Sham Comparator): Participants randomized to this group received access to an untailored general interest/lifestyle website.
  Interventions: Other: Untailored Web
- Tailored Health and Lifestyle Web (Experimental): Participants randomized to this arm received tailored web content about health and wellness, with weekly goal-setting and feedback.
  Interventions: Behavioral: Tailored Web
- Tailored Web plus Peer Coaching (Experimental): Participants randomized to this arm received access to weekly tailored health and wellness web content, plus weekly feedback from a peer health coach (videos uploaded to the web and phone calls).
  Interventions: Behavioral: Tailored Web; Behavioral: Peer Coaching

INTERVENTIONS:
Behavioral: Tailored Web — The tailored website included 6 weeks of content about making healthy lifestyle choices, eating breakfast, exercising, reducing drinking and quitting smoking. Each week, participants were asked to check in with their past week's behavior, and to set goals for the next week's check-in.
  Arms: Tailored Health and Lifestyle Web; Tailored Web plus Peer Coaching
Behavioral: Peer Coaching — Participants chose a peer coach, who reviewed the participant's check-in data and goals, and provided personalized feedback to help the participant reach those goals. Interaction took place via personalized videos recorded each week and uploaded to a participant's web profile, and through pro-active phone calls to the participants each week.
  Arms: Tailored Web plus Peer Coaching
Other: Untailored Web — Content about lifestyle issues (music, travel, dating) was created for participants assigned to the control group. There was new web content each week for 6 weeks.
  Arms: Control

SUMMARY:
The RealU2 is a randomized controlled trial to determine the efficacy of an online health and wellness program for young adults with the addition of individualized peer health coaching.

DETAILED DESCRIPTION:
The RealU addresses smoking in a young adult population of occasional and daily smokers.

Aim 1. To determine the efficacy of providing individually tailored smoking cessation messages as part of a general interest website for young adults.

Aim 2. To determine the efficacy of providing individually tailored smoking cessation messages plus peer email, phone and online support as part of a general interest website for young adults.

Participants were recruited via direct emails sent to undergraduate and graduate students at the University of MI as well as direct emails sent to participants from Survey Sampling International and National Data Group. Individuals were invited to complete an online survey about health and hope in young adults. Participants eligible for the full intervention were invited to join the RealU Study.

Participants were asked to complete an online enrollment survey and consent form. Eligible, enrolled participants were randomly assigned to one of the following three study arms:

* an untailored general interest/lifestyle website
* an individually tailored web intervention about health and lifestyle
* an individually tailored web intervention about health and lifestyle with coaching from peers, including video, phone, and email

Assessments were conducted at 7 weeks and 12 weeks post-enrollment. The primary outcome measure is self-reported 30-day abstinence at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35
* Able to read English
* Internet access for the next 3 months
* Self-reported internet use of more than once per week
* Smoked at least one puff of a cigarette in the past 30 days

Exclusion Criteria:

* Use of smokeless tobacco in the past 30 days

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1699 (Actual)
Dates: Start 2011-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Self-reported 30-day abstinence at Week 12 | 12 weeks post-enrollment
  Participants were asked how many days they had smoked in the past 30 days during the follow-up survey conducted 12-13 weeks post-enrollment.

SECONDARY OUTCOMES:
Self reported 7-day abstinence at 7 weeks | 7-weeks post-enrollment
  Participants were asked to select which of the days in the past 7 (Sun-Sat) they had smoked even one puff.
Self-reported 7-day abstinence at Week 12 | 12-weeks post-enrollment
  Participants were asked to select which days in the past 7 (Sun-Sat) they had smoked at least one puff.